CLINICAL TRIAL: NCT05912530
Title: The Influence of Gender on Dual Task Performance in Young Healthy Adults: A Cross-Sectional Study Comparing Cognitive Task and Motor Performance.
Brief Title: The Influence of Gender on Dual Task Performance in Young Healthy Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jouf University (Other)
Responsible Party: Principal Investigator, Radwa T. Elshorbagy, assistant professor, Jouf University
Other Study IDs: 2023-73
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Cognitive Change; Motor Activity
Keywords: Gender, Dual task, Cognition, Muscle torque, Speed
MeSH Terms: conditions — Motor Activity; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- male: All of the participants were Al jouf University students between the ages of 20 and 35. A BMI between 18 and 30 as well as a normal ROM at the time of the test were inclusion criteria. Additionally, participants had been excluded if they were taking any medications, showed a musculoskeletal injury to the leg, had a cognitive impairment, had a history of surgery, had a cardiovascular condition, or had any other health issue that would have an impact on their physical ability. There was no incentive for the individuals to participate. Prior to data collection, every single participant were informed that being involved in the investigation was voluntary and private, and they provided signed informed consent.
  Interventions: Other: no intervention
- female: All of the participants were Al jouf University students between the ages of 20 and 35. A BMI between 18 and 30 as well as a normal ROM at the time of the test were inclusion criteria. Additionally, participants had been excluded if they were taking any medications, showed a musculoskeletal injury to the leg, had a cognitive impairment, had a history of surgery, had a cardiovascular condition, or had any other health issue that would have an impact on their physical ability. There was no incentive for the individuals to participate. Prior to data collection, every single participant were informed that being involved in the investigation was voluntary and private, and they provided signed informed consent.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — there is no intervention will done

SUMMARY:
Dual tasking (DT), or the act of conducting multiple, simultaneous tasks, is wide spread in daily life .In particular, the vast majority of mobility tasks we complete (e.g., standing, walking, stepping, etc.) occur while distracted by another motor and/or cognitive task. A common feature of DT is that performance on one or both tasks is diminished when completed together .Understanding the relationship between gender and dual task performance is important because this knowledge could help inform us the development of interventions or training programs that target these differences and improve overall performance. Aims: To investigate the gender-related differences in single task performance through motor torque, cognitive tasks and walking speed, and the combined dual-task costs considering both motor and cognitive performance in a sample of young adults

DETAILED DESCRIPTION:
gender differences on dual task performance in young healthy adults. Dual task performance refers to the ability of an individual to perform two tasks simultaneously, which can be a challenging cognitive task because the human brain has a limited capacity for attention and processing. When an individual attempts to perform two tasks at once, they must divide their attention and resources between the two tasks, which can lead to decreased performance and increased errors.

The study will evaluate motor performance, muscle force production, and average speed through a walking test. Sixty non-athlete participants (30 female and 30 male) will be recruited, and ANCOVA will be used for statistical analysis.The participants will perform the following tasks: single mobility tasks (average speed through walking test for 45 seconds), single muscle force production, single cognitive task, dual-task condition: walking test and cognitive task, and dual-task condition: muscle torque test and cognitive task

ELIGIBILITY:
Inclusion Criteria:

* age 18-30
* BMI 18-25
* normal knee range of motion at time of test

Exclusion Criteria:

* participants had been excluded if they were taking any medications, showed a musculoskeletal injury to the leg, had a cognitive impairment, had a history of surgery, had a cardiovascular condition, or had any other health issue that would have an impact on their physical ability.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — yes
Study Population: healthy ,non athletic, young adult subjects
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Cognition | 45 seconds
  a serial subtraction of 3 from a random number between 100 and 150, the duration of each cognitive tasks was measured using a stopwatch of 45s.

SECONDARY OUTCOMES:
Average speed | 45 seconds
  One step app by iphone
Muscle force production | 45 seconds
  The Biodex System 4-Pro Isokinetic Strength Dynamometer was used to quantify muscle torque in the knee extension

CONTACTS AND LOCATIONS:
Locations (1):
- Jouf University, Sakakah, Jouf, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
study result
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after publication
Access Criteria: Study protocol